CLINICAL TRIAL: NCT06207032
Title: TEMPUS ARIES: A Biobank Registry Platform Study in Oncology
Status: Recruiting | Type: Observational
Sponsor: Tempus AI (Industry)
Responsible Party: Sponsor
Other Study IDs: TP-CA-007; Pro00076336 (Other: Advarra)
Record Dates: First submitted 2024-01-05; First posted 2024-01-16 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Cancer
Keywords: ctDNA; Next-Generation Sequencing; Oncology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood will be collected at pre-specified baseline, on-treatment and post-treatment timepoints. Left-over tissue may be collected from standard of care procedures depending on the indication.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- Cohort 001: KRAS mutated CRC: No intervention.
- Cohort 002: KRAS mutated PDAC: No intervention.
- Cohort 003: KRAS mutated NSCLC: No intervention.
- Cohort 004: Gastric 1L Plus: No intervention.
- Cohort 005: mCRPC 1L Plus: No intervention.
- Cohort 006: Pan Tumor ADCs: No intervention.

SUMMARY:
This study is a non-interventional, multicenter, multicohort evaluation of participants with cancer who will undergo longitudinal plasma ctDNA biomarker profiling at specific time points in addition to standard of care therapy.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age
2. Willing to participate in the research
3. Able to provide informed consent
4. Must be diagnosed with cancer

Exclusion Criteria:

1. Not willing or able to have additional blood samples collected

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants diagnosed with cancer willing to have additional blood samples collected for ctDNA research.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-06-26 (Actual); Primary Completion 2029-06-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Changes in ctDNA from baseline, on-treatment and post-treatment blood samples. | 5 years
  Assess ctDNA kinetics using ctDNA clearance factors such as time to clearance, best overall clearance rate, best confirmed clearance, and time to ctDNA recurrence and correlate with standard of care therapy real-world outcomes such as overall survival, progression-free survival, time to next treatment, and time to treatment discontinuation.

SECONDARY OUTCOMES:
Generation of DNA, RNA, immune and other multiomic datasets. | 5 years
  Use blood and tissue based next generation sequencing to uncover biomarkers that may predict outcomes, identify markers related to disease, identify markers related to mechanism of drug action, and inform future research.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Ting-Lin, MD, Study Director — Tempus AI, Inc.
Locations (28):
- United States (27):
  - Alabama Oncology, Birmingham, Alabama
  - PIH Health Whittier Hospital & PIH Health Physicians, Whittier, California
  - Eastern CT and Hematology and Oncology Associates, Norwich, Connecticut
  - Cancer Specialists of North Florida, Jacksonville, Florida
  - Morehouse, Atlanta, Georgia
  - Southern Illinois Healthcare, Carterville, Illinois
  - Hope and Healing Cancer Services, Hinsdale, Illinois
  - Cancer Care Specialists of Illinois, O'Fallon, Illinois
  - Illinois Cancer Care, Peoria, Illinois
  - Northwest Oncology and Hematology, Rolling Meadows, Illinois
  - Fort Wayne, Fort Wayne, Indiana
  - Goshen Center for Cancer Care, Goshen, Indiana
  - St. Claire Healthcare, Morehead, Kentucky
  - Frederick Health Regional System, Frederick, Maryland
  - Southcoast Centers for Cancer Care, Fairhaven, Massachusetts
  - Hannibal Regional Healthcare System, Inc., Hannibal, Missouri
  - Lake Regional Health, Osage Beach, Missouri
  - Oncology Hematology Associates, Springfield, Missouri
  - Hope Cancer Care of Nevada, Las Vegas, Nevada
  - Cancer Care Specialists - Reno, Reno, Nevada
  - New Jersey Cancer Center, Belleville, New Jersey
  - Regional Cancer Care Associates, Belleville, New Jersey
  - Hematology Oncology Associates of Central NY, East Syracuse, New York
  - Cayuga Medical Center, Ithaca, New York
  - Sanford Roger Maris Cancer Center (Fargo), Fargo, North Dakota
  - Taylor Cancer Research Center, Maumee, Ohio
  - Cancer Care Associates of York, York, Pennsylvania
- Pan American Center for Oncology Trials, Rio Piedras, Puerto Rico, Puerto Rico

REFERENCES:
- [Background] Thomas M. Pharma and the benefits of Real World Data. Drug Discovery World (DDW). Published November 4, 2021. Accessed May 5, 2023. https://www.ddw-online.com/trends-analysis-pharma-and-the-benefits-of-real-world-data-13702-202111/
- [Background] Office of the Commissioner. Oncology Real World Evidence Program. U.S. Food and Drug Administration. Accessed May 5, 2023. https://www.fda.gov/about-fda/oncology-center-excellence/oncology-real-world-evidence-program
- [Background] Abbosh C, Birkbak NJ, Swanton C. Early stage NSCLC - challenges to implementing ctDNA-based screening and MRD detection. Nat Rev Clin Oncol. 2018 Sep;15(9):577-586. doi: 10.1038/s41571-018-0058-3. PMID 29968853
- [Background] Vellanki PJ, Ghosh S, Pathak A, Fusco MJ, Bloomquist EW, Tang S, Singh H, Philip R, Pazdur R, Beaver JA. Regulatory implications of ctDNA in immuno-oncology for solid tumors. J Immunother Cancer. 2023 Feb;11(2):e005344. doi: 10.1136/jitc-2022-005344. PMID 36796877
- [Background] Grayson N. Real-world data can help make better drugs and do it faster. STAT. Published May 2, 2018. Accessed May 5, 2023. https://www.statnews.com/2018/05/02/real-world-data-drug-development/
- [Background] Use of circulating tumor deoxyribonucleic acid for early-stage solid tumor drug development; Draft guidance for industry. Accessed September 8, 2023. https://www.fda.gov/media/158072/
- [Background] Beaubier N, Tell R, Lau D, Parsons JR, Bush S, Perera J, Sorrells S, Baker T, Chang A, Michuda J, Iguartua C, MacNeil S, Shah K, Ellis P, Yeatts K, Mahon B, Taxter T, Bontrager M, Khan A, Huether R, Lefkofsky E, White KP. Clinical validation of the tempus xT next-generation targeted oncology sequencing assay. Oncotarget. 2019 Mar 22;10(24):2384-2396. doi: 10.18632/oncotarget.26797. eCollection 2019 Mar 22. PMID 31040929
- [Background] Beaubier N, Bontrager M, Huether R, Igartua C, Lau D, Tell R, Bobe AM, Bush S, Chang AL, Hoskinson DC, Khan AA, Kudalkar E, Leibowitz BD, Lozachmeur A, Michuda J, Parsons J, Perera JF, Salahudeen A, Shah KP, Taxter T, Zhu W, White KP. Integrated genomic profiling expands clinical options for patients with cancer. Nat Biotechnol. 2019 Nov;37(11):1351-1360. doi: 10.1038/s41587-019-0259-z. Epub 2019 Sep 30. PMID 31570899
- [Background] Finkle JD, Boulos H, Driessen TM, Lo C, Blidner RA, Hafez A, Khan AA, Lozac'hmeur A, McKinnon KE, Perera J, Zhu W, Dowlati A, White KP, Tell R, Beaubier N. Validation of a liquid biopsy assay with molecular and clinical profiling of circulating tumor DNA. NPJ Precis Oncol. 2021 Jul 2;5(1):63. doi: 10.1038/s41698-021-00202-2. PMID 34215841